CLINICAL TRIAL: NCT07158268
Title: A Phase 2 Multicenter, Randomized, Double-blind and Two-Stage Study to Evaluate the Efficacy and Safety of HSK47388 for the Treatment of Participants With Moderate to Severe Plaque Psoriasis
Brief Title: A Phase 2 Study of HSK47388 Tablets to Evaluate the Efficacy and Safety in Patients With Moderate-to-Severe Plaque Psoriasis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSK47388-201
Record Dates: First submitted 2025-08-28; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Plaque Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HSK47388 matching placebo will be administered orally. (Placebo Comparator)
  Interventions: Drug: HSK47388
- HSK47388 dose 1 will be administered orally. (Experimental)
  Interventions: Drug: HSK47388
- HSK47388 dose 2 will be administered orally. (Experimental)
  Interventions: Drug: HSK47388
- HSK47388 dose 3 will be administered orally. (Experimental)
  Interventions: Drug: HSK47388

INTERVENTIONS:
Drug: HSK47388 — HSK47388 tablets will be administered orally, once a day

SUMMARY:
The primary objective of this study is to evaluate the efficacy of multiple-dose HSK47388 versus placebo in participants with moderate-to-severe plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of plaque psoriasis with a disease duration of at least 26 weeks before the first administration of the study intervention
2. Total Body Surface Area (BSA) involvement ≥ 10% at both screening and baseline visits
3. Psoriasis Area and Severity Index (PASI) total score ≥ 12 at both screening and baseline visits
4. Investigator Global Assessment (IGA) for plaque psoriasis total score ≥ 3 (moderate or severe disease) at both screening and baseline visits
5. Participants deemed appropriate candidates for systemic therapy for plaque psoriasis

Exclusion Criteria:

1. Non-plaque psoriasis (e.g., erythrodermic, guttate, or pustular psoriasis)
2. Current drug-induced psoriasis
3. Current diagnosis, signs, or symptoms of severe, progressive, or uncontrolled disease involving the renal, hepatic, cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, or metabolic systems
4. Known allergy, hypersensitivity, or intolerance to HSK47388。
5. A history of malignant tumor before screening;
6. Subjects deemed unsuitable for participation due to other factors as determined by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-12-20 (Estimated); Study Completion 2027-01-17 (Estimated)

PRIMARY OUTCOMES:
HSK47388 and Placebo Group: Percentage of Participants Achieving PASI 75 Response From Baseline to week 16 | 16 weeks
  Percentage of participants achieving PASI 75 response (>=75% improvement in PASI from baseline) at Week 16 will be reported. The PASI is a system for assessing/grading psoriatic lesion severity and treatment response. It divides the body into 4 regions (head, trunk, upper extremities, lower extremities), with each region separately scored for erythema, induration, scaling (0-4 scale each) and involvement extent (0-6 scale). PASI yields a 0-72 numeric score, where higher scores mean more severe disease.

SECONDARY OUTCOMES:
HSK47388 and placebo Group: Percentage of Participants Achieving an IGA Score of 0 or 1 and >=2 Grade Improvement From Baseline at Weeks 16 | 16 weeks
  The percentage of participants with IGA 0/1 and ≥2-grade improvement from baseline at Weeks 16 will be reported. IGA is investigators' assessment of participants' psoriasis at a specific time point, grading overall lesions by induration, erythema, scaling, and categorizing psoriasis as cleared (0), minimal (1), mild (2), moderate (3), or severe (4).
Change From Baseline in Body Surface Area (BSA) at Week 16 | 16 weeks
  Change from baseline in BSA at Week 16 will be reported. BSA is a common measure of skin disease extent, defined as the percentage of total body surface area affected by the target condition (i.e., plaque psoriasis).
HSK47388 and Placebo Group: Change From Baseline in Total DLQI Score at Week 16 | 16 weeks
  Change from baseline in total DLQI score at Week 16 will be reported. The DLQI is a dermatology-specific HRQoL instrument designed to assess a disease's impact on participants' HRQoL. It is a 10-item questionnaire evaluating HRQoL over the past week; in addition to overall HRQoL, it assesses 6 quality-of-life domains: symptoms/feelings, daily activities, leisure, work/school performance, personal relationships, and treatment. Total scores range from 0 to 30, with higher scores indicating greater HRQoL impact.
Number of Participants with Adverse Events (AEs) | 20 weeks
  An adverse event (AE) is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.